CLINICAL TRIAL: NCT07121413
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of SV001 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of SV001 in Patients With Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Synvida Biotechnology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SV001-201
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis(IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SV001 (Experimental)
  Interventions: Drug: SV001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SV001 — SV001 ： Multiple-dose
  Arms: SV001
Drug: Placebo — Placebo ： Multiple-dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, PK and immunogenicity of SV001 in patients with idiopathic pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a confirmed diagnosis of IPF and pulmonary function meeting the protocol-specified criteria;
2. Subjects must agree to use highly effective contraception during the study and for 6 months after the last administration of the study drug;
3. Subjucts must be able to understand the study, voluntarily provide written informed consent, and be willing and able to comply with all study-related procedures.

Exclusion Criteria:

1. Subjects with a history of drug or other allergies, or those judged by the investigator to be potentially allergic to the study drugs;
2. Presence of any other clinically significant pulmonary diseases besides IPF at screening;
3. Any known contraindications to performing pulmonary function tests at screening;
4. Respiratory or systemic infections requiring anti-infective therapy within 1 month prior to randomization;
5. Acute exacerbation of IPF within 4 months prior to randomization;
6. Use of any medication known to cause or worsen pulmonary fibrosis, as assessed by the investigator, within 3 months prior to screening;
7. History of smoking within 3 months prior to screening, or unwillingness to quit smoking throughout the study period;
8. Presence of clinically significant cardiovascular, cerebrovascular, hematological, neurological, psychiatric, or metabolic disease at screening, or plans for major surgery during the study period;
9. Presence of specified abnormal laboratory test results at screening;
10. Evidence of renal impairment or end-stage renal disease requiring dialysis at screening;
11. Active hepatitis virus infection; history of acquired or congenital immunodeficiency disease;
12. History of malignancy within 5 years prior to screening;
13. Difficulty with venipuncture or a history of needle phobia or blood phobia;
14. Positive pregnancy tests or currently lactating at screening;
15. Participation in another clinical trial and receipt of other investigational drugs within 3 months prior to randomization;
16. Any other condition that the investigator consider unsuitable for participation in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 1 years
  Adverse event type, incidence, duration

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Approximately 1 years
  PK (Pharmacokinetics)
Peak time（Tmax） | Approximately 1 years
  PK (Pharmacokinetics)
Area under the plasma concentration versus time curve (AUC) | Approximately 1 years
  PK (Pharmacokinetics)
half-life（T1/2） | Approximately 1 years
  PK (Pharmacokinetics)
Immunogenicity | Approximately 1 years
  ADA（Anti-drug antibody）

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - The Affiliated Hospital of Inner Mongolia Medical University, Neimeng
  - Dongfang Hospital Affiliated to Tongji University, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - General Hospital of Tianjin Medical University, Tianjin
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Provincial People's Hospital, Zhengzhou